CLINICAL TRIAL: NCT06509685
Title: Effects of Ladder Versus Balance Training on Dynamic Balance and Performance Among Football Players
Acronym: ELVBTDBPFB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0487
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Sports Physical Therapy
Keywords: Agility; Balance exercises; Dynamic Balance; Football Players; Ladder Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): 9 participants will be in experimental group A and will perform ladder training protocol including two foot run, Ladder traps, Lateral angle leg hops, Single leg forward hop, two-foot lateral run, Fight shuffle exercises.
  Interventions: Other: Ladder Training
- Group B (Experimental): 9 participants will be in experimental group B and will perform balance training protocol including balance and landing activities incorporating wobble boards and change of direction activities
  Interventions: Other: balance training

INTERVENTIONS:
Other: Ladder Training — 9 participants will perform only Ladder training exercise protocol. The training schedule included exercises such as Two foot run, Ladder traps, Lateral angle leg hops, Single leg forward hop, two-foot lateral run, Fight shuffle, Skiers, Carioca, Lateral in out, two in two out, Intermediate high knee run, Straddle squat hops, two foot laterals hop in & out, Two-foot lateral hop, Ali shuffle, 180 Degree rotation, jumping jacks' variation, Advanced in in out, Quick hops cotch, Icky shuffle etc. For each session, ten stations were used and participants change the partner after every end of steps jumping exercise and continued each exercise at least 3 set, depending on the class design(22).
  Arms: Group A
Other: balance training — 9 participants will perform balance training protocol. The balance training program includes exercises based around balance development in unilateral dynamic balancing positions. The program included balance and landing activities incorporating wobble boards and change of direction activities.
  Arms: Group B

SUMMARY:
Football is becoming more and more popular around the world since it is easier to obtain. Depending on specific game activities, a player's position on the field may have an impact on their physical traits. Ladder and Balance training is a well-recognized technique for improving players' multidirectional footwork and dynamic balance-both crucial for the rigorous demands of football. The objective of this study is to determine the effects of ladder versus balance training on dynamic balance and performance of football players.

The study design is Randomized Clinical Trial (RCT). The sample size was calculated from epitool software. This study would include total n= 20 participants which would be divided equally into Group A- ladder Training (n=9) and Group B-balance Training (n=9). The study will be conducted in Bahria Football Academy. Modified Star Excursion Balance Test (SEBT) assesses dynamic balance while performance include Vertical Jump, Dribbling, 30m Sprint, and Illinois Agility evaluation at baseline and after 6th-weeks. The data will be analyzed using SPSS version 28.

DETAILED DESCRIPTION:
This study investigates the comparative effects of ladder training and balance training on dynamic balance and performance in football players. The research aims to understand how these distinct training modalities impact dynamic balance and overall performance, providing valuable insights for coaches and athletes. The goal is to tailor training regimens to optimize specific athletic aspects essential in football, contributing to the evidence base for designing more effective protocols in football player development.

ELIGIBILITY:
Inclusion Criteria:

* Male Football Players
* Age 18 to 25 Years
* Participants who regularly trained in football
* Participants who were from various amateur football teams participated in the study

Exclusion Criteria:

* Participants who had an injury in the previous six months
* Participants who underwent any surgery with in last one year
* Participants were excluded if they reported any current injury that limited daily activity

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 18 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Modified Star Excursion Balance Test (SEBT) | 8 weeks
  Star excursion balance test in the earlier days include 8 reach directions. Participants reported for a single testing session. The dominant leg will be determined as the leg used by the participant for kicking. The length of both the legs will be measured from the anterior superior iliac spine to the middle of the medial malleolus using a standard tape measure while participants lay supine on a plinth. The task goal and performance constraints of the SEBT will be explained to the participants. Reach directions will be evaluated by affixing three tape measures to the floor, one orientated anterior to the apex (A) and two aligned at 135 to this in the Posteromedial and Posterolateral directions.
Vertical Jump test | 8 weeks
  The person stands side on to a wall and reaches up with the hand closest to the wall. Keeping the feet flat on the ground, the point of the fingertips is marked or recorded. The person puts chalk on their fingertips to mark the wall at the height of their jump. The person then stands away from the wall and jumps vertically as high as possible using both arms and legs to assist in projecting the body upwards. Attempt to touch the wall at the highest point of the jump.
30-m sprint test | 8 weeks
  The test involves running a single maximum sprint over 30 meters, with the time recorded. A thorough warm up should be given, including some practice starts and accelerations. Start from a stationary position, with one foot in front of the other. The front foot must be on or behind the starting line. This starting position should be held for 2 seconds prior to starting, and no rocking movements are allowed. The tester should provide hints for maximizing speed (such as keeping low, driving hard with the arms and legs) and encourage them to continue running hard through the finish line.
Illinois Agility Test | 8 weeks
  The individual starts by lying face down by the first cone. Staring at cone 1 he is required to run to cone 2 which is placed at a distance of 10 meters away from the first. He then runs 10 meters to cone 3. At this point the individual has to weave around cones 3,4,5,6. After this he has to go through 5,4,3. He will then run to cone # 8. The time to complete the task is then recorded.
Figure 8 dribbling test | 8 weeks
  The player starts on one side of the first cone. Player must dribble around each cone in a figure8 pattern, without touching the cone, using both feet and trying to use both the inside and outside of her feet. She may also use the sole of her feet

CONTACTS AND LOCATIONS:
Overall Officials: Muzna Munir, Ph.D, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Padron-Cabo A, Rey E, Kalen A, Costa PB. Effects of Training with an Agility Ladder on Sprint, Agility, and Dribbling Performance in Youth Soccer Players. J Hum Kinet. 2020 Jul 21;73:219-228. doi: 10.2478/hukin-2019-0146. eCollection 2020 Jul. PMID 32774553
- [Background] Ksiazek A, Zagrodna A, Slowinska-Lisowska M. Assessment of the Dietary Intake of High-Rank Professional Male Football Players during a Preseason Training Week. Int J Environ Res Public Health. 2020 Nov 18;17(22):8567. doi: 10.3390/ijerph17228567. PMID 33218191
- [Background] Doganay M, Bingul BM, Alvarez-Garcia C. Effect of core training on speed, quickness and agility in young male football players. J Sports Med Phys Fitness. 2020 Sep;60(9):1240-1246. doi: 10.23736/S0022-4707.20.10999-X. PMID 33124789
- [Background] Teixeira JE, Alves AR, Ferraz R, Forte P, Leal M, Ribeiro J, Silva AJ, Barbosa TM, Monteiro AM. Effects of Chronological Age, Relative Age, and Maturation Status on Accumulated Training Load and Perceived Exertion in Young Sub-Elite Football Players. Front Physiol. 2022 Mar 31;13:832202. doi: 10.3389/fphys.2022.832202. eCollection 2022. PMID 35432006
- [Background] Beato M, Bianchi M, Coratella G, Merlini M, Drust B. Effects of Plyometric and Directional Training on Speed and Jump Performance in Elite Youth Soccer Players. J Strength Cond Res. 2018 Feb;32(2):289-296. doi: 10.1519/JSC.0000000000002371. PMID 29176387
- [Background] Saez de Villarreal E, Suarez-Arrones L, Requena B, Haff GG, Ferrete C. Effects of Plyometric and Sprint Training on Physical and Technical Skill Performance in Adolescent Soccer Players. J Strength Cond Res. 2015 Jul;29(7):1894-903. doi: 10.1519/JSC.0000000000000838. PMID 25635606
- [Background] Bedoya AA, Miltenberger MR, Lopez RM. Plyometric Training Effects on Athletic Performance in Youth Soccer Athletes: A Systematic Review. J Strength Cond Res. 2015 Aug;29(8):2351-60. doi: 10.1519/JSC.0000000000000877. PMID 25756326
- [Background] Sheppard JM, Young WB. Agility literature review: classifications, training and testing. J Sports Sci. 2006 Sep;24(9):919-32. doi: 10.1080/02640410500457109. PMID 16882626
- [Background] Michailidis Y, Fatouros IG, Primpa E, Michailidis C, Avloniti A, Chatzinikolaou A, Barbero-Alvarez JC, Tsoukas D, Douroudos II, Draganidis D, Leontsini D, Margonis K, Berberidou F, Kambas A. Plyometrics' trainability in preadolescent soccer athletes. J Strength Cond Res. 2013 Jan;27(1):38-49. doi: 10.1519/JSC.0b013e3182541ec6. PMID 22450257
- [Background] Kenville R, Maudrich T, Korner S, Zimmer J, Ragert P. Effects of Short-Term Dynamic Balance Training on Postural Stability in School-Aged Football Players and Gymnasts. Front Psychol. 2021 Nov 17;12:767036. doi: 10.3389/fpsyg.2021.767036. eCollection 2021. PMID 34867668